CLINICAL TRIAL: NCT04680520
Title: A Randomised Controlled Trial to Determine Whether Application of Emollient From Birth Can Prevent Eczema in High Risk Children.
Brief Title: Barrier Enhancement for Eczema Prevention
Acronym: BEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14044
Record Dates: First submitted 2015-12-08; First posted 2020-12-23 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Eczema
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Best practice skin care advice booklet plus emollient (Doublebase Gel® or Diprobase Cream®) (Experimental): Use of emollient (Doublebase Gel® or Diprobase Cream®) plus best practice skin care advice. The advice is given in the form of a booklet containing advice on skin care. This will contain information on avoiding soap etc. It will also explain how to apply the emollient i.e. in the direction of the hair, all over the child's skin daily for the first year of life. Intervention group will receive both emollients and parents are asked to choose their preferred.
  Interventions: Other: Experimental (Doublebase Gel® or Diprobase Cream®); Other: Best practice skin care advice booklet
- Best practice skin care advice booklet (Active Comparator): This is a booklet containing advice on best practice skin care. This will contain information on avoiding soap etc.
  Interventions: Other: Best practice skin care advice booklet

INTERVENTIONS:
Other: Experimental (Doublebase Gel® or Diprobase Cream®) — Emollient (Doublebase Gel® or Diprobase Cream®) use on the skin. The emollient should be applied at least once a day.
  Arms: Best practice skin care advice booklet plus emollient (Doublebase Gel® or Diprobase Cream®)
Other: Best practice skin care advice booklet — This is a booklet containing advice on best practice skin care. This will contain information on avoiding soap etc.

SUMMARY:
The primary objective is to determine whether advising parents to apply emollient (moisturiser) to their child's skin for the first year of life in addition to best practice infant skin care advice can prevent or delay the onset of eczema in high-risk children, when compared with a control group who are given the best practice infant skin care advice only.

ELIGIBILITY:
Inclusion Criteria:

* child has a first degree relative with parental reported doctor diagnosis of eczema, allergic rhinitis or asthma
* child up to 21 days old
* consenting adult has the ability to understand English

Exclusion Criteria:

* preterm birth (defined as birth prior to 37 weeks gestation)
* sibling (including twin) previously randomized to this trial. If multiple births, the first child will be randomized into the trial.
* child has a severe widespread skin condition that would make the detection and/or assessment or eczema difficult
* child has a serious health issue, which, at parent or investigator discretion, would make it difficult for the family to take part in the trial
* any condition that would make the use of emollient inadvisable or not possible

Max Age: 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1394 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
A diagnosis of eczema between 12 and 24 months of age (defined as meeting the United Kingdom (UK) Working Party Diagnostic Criteria for Atopic Dermatitis). | 24 months
  To reflect the chronicity of eczema, these criteria refer to signs and symptoms present over the past year. Applying the criteria at 24 months of age will therefore detect eczema present only between the ages of 12 and 24 months, thus excluding transient eczematous rashes which are common in the first year of life and often reported by parents as "eczema" but less likely to be true atopic eczema

SECONDARY OUTCOMES:
Presence of parental report of eczema between birth and 24 months. | Up to 24 months
  Assessed using:
  Any parental report of a clinical diagnosis of eczema. Completion by parents of UK Working Party Diagnostic Criteria for Atopic Dermatitis at 12 and 24 months.
Presence of visible eczema at 24 months (skin examination by researcher). | 24 months
  Presence of visible eczema at 24 months (skin examination by researcher).
Time to onset of eczema | 24 months
  First parental report of a clinical diagnosis of eczema. First topical corticosteroid and /or immunosuppressant prescription for eczema.
Presence of other allergic diseases using parental reports, allergic sensitization and confirmed diagnosis | Upto 24 months
  Parental reported wheezing and allergic rhinitis between 12 and 24 months. Parental report of a clinical diagnosis of food allergy at 12 and 24 months. Parental report of food allergy at 12 and 24 months. Parents will be specifically questioned about cow's milk, egg, peanuts, and other nuts plus "any other food".
  Allergic sensitisation at 24 months to any of the following common allergens: milk, egg, peanut, cat, grass pollen, house dust mite.
  Confirmed diagnosis of food allergy at 24 months to milk, egg, peanut or 'any of milk, egg or peanut'. The diagnosis is derived from a combination of parental report, allergic sensitisation and food challenge.
Child health-related quality adjusted life years. | Upto 24 months
  Child health utility 9 dimension (CHU-9D) at 24 months in order to estimate quality adjusted life years (QALYs).
Parental health-related quality adjusted life years. | Upto 24 months
  Parental quality of life measured using the EQ-5D-5L at baseline and 24 months in order to estimate change in parental QALYs, if any.
Cost or treatments- health economic outcomes | Up to 24 months
  Health care resource use at 3, 6, 12, 18 and 24 months. Cost effectiveness and cost-utility at 24 months (combining health resource use and health-related quality of life outcomes).
Severity of eczema with EASI eczema severity scales | Up to 24 months
  Assessed using eczema area and severity index (EASI) at 24 months. The area score is recorded for each of four regions of the body: head and neck, trunk, upper limbs and lower limbs. The area score is the percentage of skin affected by eczema for each body region. The scores given are from 0-6 where a score of 0 is given when the percentage of skin affected by eczema in the region is 0%, and a score of 6 is given when 90-100% of the region is affected by eczema. The severity score is recorded for each of the four body regions for four signs: redness, thickness, scratching and lichenification. Scores are given from 0-3 where a score of 3 is for most severe signs.
Severity of eczema with POEM eczema severity scales | Up to 24 months
  Assessed using patient oriented eczema measure (POEM) at 12 and 24 months. The scores given are from 0-28, where a score of 28 is for the most severe.

OTHER OUTCOMES:
Presence of eczema in the previous year at 36, 48 and 60 months based on parental report of a clinical diagnosis of eczema | 36, 48 and 60 months
  Presence of eczema in the previous year at 36, 48 and 60 months based on parental report of a clinical diagnosis of eczema
Any parental report that in their opinion their child has eczema at 3, 6, 12, 24, 36, 48 and 60 months | 3, 6, 12, 24, 36, 48 and 60 months
  Any parental report that in their opinion their child has eczema at 3, 6, 12, 24, 36, 48 and 60 months
Presence of eczema at 36, 48 and 60 months based on completion by parents of UK Working Party Diagnostic Criteria for Atopic Dermatitis | 36, 48 and 60 months
  Presence of eczema at 36, 48 and 60 months based on completion by parents of UK Working Party Diagnostic Criteria for Atopic Dermatitis
Severity of eczema at 36, 48, and 60 months as measured by POEM | 36, 48, and 60 months
  Severity of eczema at 36, 48, and 60 months as measured by Patient Oriented Eczema Measure (POEM)
Parental reported wheezing, at 36, 48 and 60 months | 36, 48 and 60 months
  Parental reported wheezing, at 36, 48 and 60 months
Parental reported allergic rhinitis at 36, 48 and 60 months | 36, 48 and 60 months
  Parental reported allergic rhinitis at 36, 48 and 60 months
Parental reported food allergy symptoms at 36, 48 and 60 months | 36, 48 and 60 months
  Parental reported food allergy symptoms at 36, 48 and 60 months
Parental report of a clinical diagnosis of asthma or allergic rhinitis by 60 months | By 60 months
  Parental report of a clinical diagnosis of asthma or allergic rhinitis by 60 months
Parental report of a clinical diagnosis of food allergy at 36, 48 and 60 months | 36, 48 and 60 months
  Parental report of a clinical diagnosis of food allergy at 36, 48 and 60 months
CHU-9D at 36, 48 and 60 months in order to estimate QALYs | 36, 48 and 60 months
  Child health utility 9 dimension (CHU-9D) at 36, 48 and 60 months in order to estimate quality adjusted life years (QALYs)
Parental quality of life measured using EQ-5D-5L at 36, 48 and 60 months in order to estimate parental QALYs | 36, 48 and 60 months
  Parental quality of life measured using EQ-5D-5L at 36, 48 and 60 months in order to estimate parental quality adjusted life years (QALYs)
Health care resource use at 36, 48 and 60 months | 36, 48 and 60 months
  Health care resource use at 36, 48 and 60 months
Cost utility and cost-effectiveness at 60 months (combining health resource use and health-related quality of life outcomes) | 60 months
  Cost utility and cost-effectiveness at 60 months (combining health resource use and health-related quality of life outcomes)
Parental report of clinical diagnosis of eczema from the age of 12 months to 60 months | 12 months to 60 months
  Parental report of clinical diagnosis of eczema from the age of 12 months to 60 months
Parental report of clinical diagnosis of food allergy by 60 months | By 60 months
  Parental report of clinical diagnosis of food allergy by 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Hywel Williams, Principal Investigator — Centre of Evidence-Based Dermatology, University of Nottingham.
Locations (16):
- United Kingdom (16):
  - School of Social and Community Medicine, University of Bristol, Bristol
  - Queens Hospital, Burton
  - Derby Childrens Hosptia, Derby
  - Harrogate District Hospital, Harrogate
  - Leicester Royal Infirmary, Leicester
  - Clapham Park Group Practice, London
  - Francis Grove Medical Practice, London
  - Park Group Practice, London
  - St John's Institute of Dermatology, London
  - St Mary's Hospital, London
  - Streatham Common Medical Practice, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - St Mary's Hospital, Portsmouth
  - Academic Unit of Dermatology Research, Univeristy of Sheffield, Sheffield
  - Kings Mill Hospital, Sutton in Ashfield
  - York Hospital, York

REFERENCES:
- [Result] Bradshaw LE, Wyatt LA, Brown SJ, Haines RH, Montgomery AA, Perkin MR, Lawton S, Sach TH, Chalmers JR, Ridd MJ, Flohr C, Brooks J, Swinden R, Mitchell EJ, Tarr S, Jay N, Thomas KS, Allen H, Cork MJ, Kelleher MM, Simpson EL, Lartey ST, Davies-Jones S, Boyle RJ, Williams HC. Emollients for prevention of atopic dermatitis: 5-year findings from the BEEP randomized trial. Allergy. 2023 Apr;78(4):995-1006. doi: 10.1111/all.15555. Epub 2022 Nov 3. PMID 36263451
- [Result] Chalmers JR, Haines RH, Bradshaw LE, Montgomery AA, Thomas KS, Brown SJ, Ridd MJ, Lawton S, Simpson EL, Cork MJ, Sach TH, Flohr C, Mitchell EJ, Swinden R, Tarr S, Davies-Jones S, Jay N, Kelleher MM, Perkin MR, Boyle RJ, Williams HC; BEEP study team. Daily emollient during infancy for prevention of eczema: the BEEP randomised controlled trial. Lancet. 2020 Mar 21;395(10228):962-972. doi: 10.1016/S0140-6736(19)32984-8. Epub 2020 Feb 19. PMID 32087126
- [Result] Bradshaw LE, Montgomery AA, Williams HC, Chalmers JR, Haines RH. Two-by-two factorial randomised study within a trial (SWAT) to evaluate strategies for follow-up in a randomised prevention trial. Trials. 2020 Jun 8;21(1):529. doi: 10.1186/s13063-020-04373-4. PMID 32546180